CLINICAL TRIAL: NCT00240630
Title: A Randomized, Double-blind, Multi-center, Placebo-controlled, Cross-over Study to Determine the Consistency of Response for Trexima (Sumatriptan 85mg/Naproxen Sodium 500mg) Administered During the Mild Pain Phase for the Acute Treatment of Multiple Migraine Attacks
Brief Title: Treximet (Sumatriptan/Naproxen Sodium), Formerly Known as Trexima, In The Acute Treatment Of Multiple Migraine Attacks
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TRX103632
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Migraine Disorders; Migraine
Keywords: acute migraine; consistency of response; satisfaction; migraine; early intervention
MeSH Terms: conditions — Migraine Disorders; Personal Satisfaction | interventions — Sumatriptan; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm 1 (Placebo Comparator): placebo to match
  Interventions: Drug: sumatriptan succinate/naproxen sodium
- Arm 2 (Experimental): Treximet (sumatriptan/naproxen sodium)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sumatriptan succinate/naproxen sodium — Combination Tablet of Treximet
  Arms: Arm 1
Drug: placebo — placebo to match
  Arms: Arm 2

SUMMARY:
The purpose of this study is to determine the consistency of response for Treximet (sumatriptan/naproxen sodium), formerly known as Trexima, when treating four acute migraine attacks at the mild pain phase and within 1 hour of onset of head pain.

ELIGIBILITY:
Inclusion Criteria:

* At least a 6 month history of physician diagnosed migraine and typically experiences 2-6 migraine attacks per month.
* Typically experiences moderate to severe migraine pain preceded by a mild pain phase.
* Differentiate between mild migraine pain and other headache types.
* Women of childbearing potential must be on adequate contraception.

Exclusion Criteria:

* Pregnant and/or nursing mother.
* History of cardiovascular disease.
* Uncontrolled hypertension.
* Basilar or Hemiplegic migraine.
* History of stroke or transient ischemic attacks (TIA).
* History of epilepsy or treated with anti-epileptics within past 5 years.
* Impaired hepatic or renal function.
* History of gastrointestinal bleeding or ulceration.
* Allergy or hypersensitivity to Aspirin or any other NSAID.
* Allergy or hypersensitivity to triptans.
* Participated in an investigational drug trial in the previous 4 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2005-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Score on a migraine pain scale for multiple migraine attacks | 2 to 24 hours

SECONDARY OUTCOMES:
Within patient consistency of response, freedom from all migraine pain and symptoms, satisfaction, presence or absence of neck pain/discomfort, sinus pain/pressure, recurrence of head pain, safety and tolerability | 2 to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (48):
- United States (48):
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Westlake Village, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Palm Beach Gardens, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Austell, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Braintree, Massachusetts
  - GSK Investigational Site, Milford, Massachusetts
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Endwell, New York
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, Manlius, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Georgetown, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Burlington, Vermont
  - GSK Investigational Site, Seattle, Washington

REFERENCES:
- [Result] Torgovnick J, Sethi NK, Arsura E. Consistency of response to sumatriptan/naproxen sodium in a placebo-controlled cross-over study. Cephalalgia. 2010 Oct;30(10):1277; author reply 1277-9. doi: 10.1177/0333102409352810. Epub 2010 May 13. No abstract available. PMID 20855373